CLINICAL TRIAL: NCT03232528
Title: A Study on the Promotion Plan of the Moxibustion Treatment of Ulcerate Colitis
Brief Title: The Promotion Plan of Moxibustion on Ulcerate Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: promotion
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Herb-partitioned moxibustion (Experimental): Drug: Herbal cake, Device: Moxibustion. Herbal cakes formula: Monkshood 10g, Cinnamon 2g, Salvia miltiorrhiza 3g, Flos Carthami 3g, Radix Aucklandiae 2g. Herbs are smashed into powder. Every 2.5g medicine powder is mixed with 3g millet wine and then pressed into herbal cakes using a specific mold. Each cake should be 23mm in diameter and 5mm in height. Then, ignited moxa cones are placed on top of each herbal cake. Herbal cakes with moxa cones will be positioned at acupuncture points ST25, ST37 and CV6. The entire treatment will be done once a day for 1 moxa cone every acupuncture point, 30 minutes at a time, 3 times a week, for a total of 12 weeks.
  Interventions: Other: Herb-partitioned moxibustion
- Sham herb-partitioned moxibustion (Sham Comparator): Drug: Herbal cake, Device: Sham moxibustion. Herbal cakes formula: Monkshood 10g, Cinnamon 2g, Salvia miltiorrhiza 3g, Flos Carthami 3g, Radix Aucklandiae 2g. Herbs are smashed into powder. Every 2.5g medicine powder is mixed with 3g millet wine and then pressed into herbal cakes using a specific mold. Each cake should be 23mm in diameter and 5mm in height. Then, ignited moxa cones are placed on top of each herbal cake. Small cardboard sheets with the same size as the herbal cakes will be wrapped with aluminum foil and placed under each herbal cake. These herbal cakes will be positioned at acupuncture points ST25, ST37 and CV6. The entire treatment will be done once a day for 1 moxa cone every acupuncture point, 30 minutes at a time, 3 times a week, for a total of 12 weeks.
  Interventions: Other: Sham herb-partitioned moxibustion

INTERVENTIONS:
Other: Herb-partitioned moxibustion — Patients receive herb-partition moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks.
  Other Names: Treatment Group
  Arms: Herb-partitioned moxibustion
Other: Sham herb-partitioned moxibustion — Patients receive sham herb-partition moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks.
  Other Names: Control Group
  Arms: Sham herb-partitioned moxibustion

SUMMARY:
To evaluate the efficacy of Moxibustion in the treatment of Ulcerative Colitis, thus the scientific foundation for rational use of Moxibustion in clinical usage, in order to find admission of the Acupuncture and Moxibustion and even medicine field, accomplish popularization and application.

DETAILED DESCRIPTION:
A total of 128 patients with UC were randomly divided into the following 2 groups: a) Herb-partition moxibustion (Treatment Group) and b) Sham herb-partition moxibustion (Control Group). All patients in the trial will be treated with moxibustion 3 times a week, once a day for 30 minutes, for a total of 12 weeks. After treating the treatment had ended and the 52nd week of follow-up to observe the clinical therapy effect of Moxibustion in UC patients. Tissue morphology and molecular biology tests will be conducted to observe the regulation in the intestinal mucosa of UC patients. All these steps will be done in order to provide clinical usage for the effects of herb-partition moxibustion in the treatment of UC.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnosis of UC
* Patients do not receive any medicine, or if they are receiving medicine, it should be aminosalicylates and/or prednisone (dose ≤15mg and have taken at least 1 month);
* Patients should have not received antibiotic, biologicals within 3 months prior to entering the study;
* Signing a written informed consent.

Exclusion Criteria:

* Patients with cardiac, encephalic, hepatic, nephric, hematopoietic system, psychotic or any other serious diseases;
* Pregnancy or lactation;
* genetic family history of nervous system disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
total effective rate | 3 months
  The curative effect of Herb-partitioned moxibustion for 128 UC patients.

SECONDARY OUTCOMES:
Mayo score | 6 months
  Assay for the ulcerative colitis desease activity index. It is constructed by four scales, Including stool frequency、rectal bleeding、mucosal appearance at endoscopy and physician rating of disease activity. Every scale can be scored with o ,1 ,2 or 3 according to the activity index of scale. Scores should be compared to previous scores taken for a patient. The higher the score (minimum 0 point and maximum 12 points), the more severe the ulcerative colitis.
symptom score | 3 months
  Observe the abdominal pain, bloody stool, intolerance of cold, soreness and weakness of waist an knees, diarrhea, mucous stool, tenesmus, anorexia and lassitude score.
Visual Analogue Scale(VAS) | 6 months
  Observe the degree of abdominal pain
Inflammatory Bowel Disease Questionnaire(IBDQ) | 6 months
  Life quality was determined by the total score of the 32 questions. Each question is given 1-7 different degrees of answer. One represents the heaviest degree and seven represents the lightest degree. The lower the score (minimum 32 points and maximum 224 points), the worse the life quality.
Hospital Anxiety and Depression Scale(HADS) | 3 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 .The higher the total score (minimum 0 point and maximum 21 points), the more severe the anxiety or depression.
Laboratory tests for disease activity: C-reaction protein | 6 months
  Assay for the quantification of total C-reaction protein in serum.(Normal reference value:<10mg/L)
Laboratory tests for disease activity: Erythrocyte sedimentation rate | 6 months
  Assay for the quantification of total Erythrocyte sedimentation rate in serum.(Normal reference value: male 0～15mm/h; female 0～20mm/h)
gut mucosal score under the endoscopy: Baron score; | 3 months
  evaluate the gut mucosal state by using electronic colonoscopy
mucosal pathology：Geboes score | 3 months
  Observe the intestinal mucosal tissue changes by HE staining

OTHER OUTCOMES:
Safety Assessment | 3 months
  With Administration Events reports record the adverse reaction treatment process, with the moxibustion treatment of safety evaluation. Such as the incidence and severity of scald, skin allergic, vasodepressor syncope etc. Also record subjects's vital signs, consist of body temperature, blood pressure and pulse.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, Doctor, Study Director — Shanghai Institute of Acupuncture-Moxibustion and Meridian, Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai Research Insititute of Acupuncture and Meridian, Shanghai, Xuhui, China